CLINICAL TRIAL: NCT04905303
Title: Prospective Multi-center, Single-arm Registry to Evaluate the Efficacy of the Solitaire AB Neurovascular Remodeling Device in the Treatment of Wide-neck Intracranial Aneurysms
Brief Title: Solitaire Aneurysm Remodeling Registry
Status: Withdrawn | Type: Observational
Sponsor: Medtronic Neurovascular Clinical Affairs (Industry)
Responsible Party: Sponsor
Other Study IDs: SOLARE
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Intracranial Saccular Aneurysm, Either Rupture or Unruptured; Wide Neck Aneurysm
Keywords: Intracranial aneurysms; Wide neck aneurysms
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of the registry is to evaluate the effectiveness and performance of the Solitaire Neurovascular Remodeling Device when used with embolic coils in the treatment of intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of intracranial saccular aneurysms, either ruptured or unruptured
* Aneurysm requires current treatment with coils and a stent or aneurysm hs been previously treated with coils, but no prior placement of a stent.
* Aneurysm has a wide neck defined as having a neck equal to or greater than 4mm or a dome-to-neck ratio of <2.
* Patient is 18 years or older.
* Patient has a Hunt & Hess score of III or less.

Exclusion Criteria:

* Patient has a fusiform or dissecting aneurysm type.
* Patient is contraindicated for either heparin or anti-platelet therapy.
* Patient has severe allergy to IV contrast medium.
* Patient has a known hypersensitivity to nickel-titanium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed diagnosis of intracranial saccular aneurysm which can be treated with coil embolization and neurovascular stenting.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2011-02 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Stable Stent placement with complete coverage across the aneurysm neck with parent artery patency | Six months post-implant

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Neurologique, Lyon, France